CLINICAL TRIAL: NCT01050777
Title: Pilot Study of Efficacy of Topical Nano-liposomal Meglumine Antimoniate (Glucantime) or Paromomycin in Combination With Systemic Glucantime for the Treatment of Anthroponotic Cutaneous Leishmaniasis (ACL) Caused by Leishmania Tropica
Brief Title: Efficacy of Topical Liposomal Form of Drugs in Cutaneous Leishmaniasis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Mashhad University of Medical Sciences (Other); Center for Research and Training in Skin Diseases and Leprosy (Unknown)
Responsible Party: Principal Investigator, Ali Khamesipour, PhD, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 86783
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2011-02

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous Leishmaniasis caused by l. tropica
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Liposomal Paromomycin (Experimental): Liposomes containing 10% Paromomycin
  Interventions: Drug: Liposomal meglumine antimoniate; Drug: Liposomal Paromomycin
- Liposomal meglumine antimoniate (Experimental): Liposomes containing meglumine antimonate
  Interventions: Drug: Liposomal meglumine antimoniate (Glucantime); Drug: Liposomal meglumine antimoniate
- Placebo (Placebo Comparator)
  Interventions: Drug: Liposomal meglumine antimoniate; Drug: Placebo

INTERVENTIONS:
Drug: Liposomal meglumine antimoniate (Glucantime) — Liposomes containing meglumine antimoniate
  Arms: Liposomal meglumine antimoniate
Drug: Liposomal meglumine antimoniate — Liposomal form of meglumine antimoniate
Drug: Liposomal Paromomycin — Liposomal form of 10% Paromomycin
  Arms: Liposomal Paromomycin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Leishmaniasis with diverse clinical manifestations is caused by different species of Leishmania and is endemic in many countries. Although Cutaneous Leishmaniasis (CL) is a self-healing disease, but it takes a long time to heal. Pentavalent antimonials are still the first-line treatment of CL which needs multiple injections, are painful and as such not tolerated by most of the patients, in addition available treatments are not always effective and resistance is reported. Paromomycin sulfate (PM) reported to show anti-Leishmania activity against both CL and visceral leishmaniasis (VL) since 1960s. Therapeutic strategy with high efficacy is urgently needed especially for Anthroponotic Cutaneous Leishmaniasis (ACL). Liposomes are lipid bilayer molecules which entrap water-soluble molecules in their internal water compartment and water-insoluble ones into their lipid bilayers. Liposomes, in proper formulations and sizes, deliver drugs to the skin based on the similarity of the bilayers structure of lipid vesicles to that of natural membrane and target the macrophages within dermis. Several lipid-based formulations have been developed to treat experimental leishmaniasis. Recently different doses of liposomal formulation of PM and liposomal formulation of Glucantime were prepared and showed high efficacy in vivo against L. major infection in BALB/c mice.

In this study the efficacy of liposomal formulation of PM or liposomal formulation of Glucantime in combination with systemic Glucantime in the treatment of ACL parasitologically proven patients will be evaluated. The clinical trial will be carried out according to the International approved GCP (Good Clinical Practice) guide lines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 12 to 60 years.
* Parasitologically proven CL due to L. tropica.
* History of failure to at least one full course of systemic Glucantime.
* In general good health based on history and physical examination.
* Number of lesion at most 4.
* Lesion size less than 3 cm.
* Signed informed consent voluntarily and knowingly.

  * Guardian's signature for volunteer less than 18 years old.

Exclusion Criteria:

* Pregnant or lactating women and those who are planning to be pregnant in next 60 days.
* Use of other types of treatment for CL.
* Involvement in any other drug or vaccine trial during the study period.
* Known heart, kidney, liver diseases based on history and physical exam. Abnormal ECG.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Complete cure equal to Complete Re-epithelization of all lesions | 200 days

CONTACTS AND LOCATIONS:
Overall Officials: Masud Maleki, MD, Principal Investigator — Mashhad University of Medical Sciences, Mashhad, Iran; Ali Khamesipour, MPH, PhD, Principal Investigator — Center for Research & Training in Skin Diseases & Leprosy, TUMS; Mahmoud Reza Jaafari, Parm D, PhD, Principal Investigator — Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Emam Reza Hospital, Mashhad, Khorasan Razavi, Iran